CLINICAL TRIAL: NCT06411860
Title: A Randomized, Placebo- and Positive-controlled, Crossover Study to Assess the Effect of Olpasiran (AMG 890) on QT/QTc Intervals in Healthy Subjects
Brief Title: A Study to Assess the Effect of Olpasiran on QT/QTc Intervals in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 20220016
Record Dates: First submitted 2024-04-29; First posted 2024-05-13 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Basic Science
Keywords: QT/QTc Intervals; Healthy Participants; Olpasiran; AMG 890
MeSH Terms: interventions — olpasiran; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A (Placebo Comparator): All participants will be randomized to 1 of 12 treatment sequences and receive a single dose of one of the following treatments, according to the randomization schedule:
  Treatment A: placebo Treatment B: dose level 1 olpasiran Treatment C: dose level 2 olpasiran Treatment D: moxifloxacin
  Interventions: Other: Placebo
- Treatment B (Experimental): All participants will be randomized to 1 of 12 treatment sequences and receive a single dose of one of the following treatments, according to the randomization schedule:
  Treatment A: placebo Treatment B: dose level 1 olpasiran Treatment C: dose level 2 olpasiran Treatment D: moxifloxacin
  Interventions: Drug: Olpasiran
- Treatment C (Experimental): All participants will be randomized to 1 of 12 treatment sequences and receive a single dose of one of the following treatments, according to the randomization schedule:
  Treatment A: placebo Treatment B: dose level 1 olpasiran Treatment C: dose level 2 olpasiran Treatment D: moxifloxacin
  Interventions: Drug: Olpasiran
- Treatment D (Active Comparator): All participants will be randomized to 1 of 12 treatment sequences and receive a single dose of one of the following treatments, according to the randomization schedule:
  Treatment A: placebo Treatment B: dose level 1 olpasiran Treatment C: dose level 2 olpasiran Treatment D: moxifloxacin
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Other: Placebo — Participants will receive a subcutaneous (SC) injection of placebo.
  Arms: Treatment A
Drug: Olpasiran — Participants will receive a SC injection of olpasiran at dose level 1 or 2.
  Arms: Treatment B; Treatment C
Drug: Moxifloxacin — Participants will receive a single dose of moxifloxacin as an oral tablet by mouth.
  Arms: Treatment D

SUMMARY:
The primary objective of the study is:

• To assess the effects of a single therapeutic and supratherapeutic dose of olpasiran on the placebo-corrected change from baseline in QT corrected for heart rate (ΔΔQT)/QTc interval in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent prior to starting study activities.
* Healthy male or female participants, between 18 and 60 years of age (inclusive) at the time of Screening. Females must be of nonchildbearing potential.
* Body mass index between 18 and 30 kg/m^2 (inclusive) at the time of Screening. Participants must have a body mass ≥ 50kg.

Exclusion Criteria:

* History or evidence, at Screening or Check-in, of clinically significant disorder, condition, or disease not otherwise excluded that, in the opinion of the Investigator (or designee), would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion.
* History or current signs or symptoms of cardiovascular disease, including but not limited to myocardial infarction, congenital heart disease, valvular heart disease coronary revascularization, or angina.
* History or evidence of clinically significant arrhythmia at screening, including any clinically significant findings on the ECG taken at Check-in.
* Systolic blood pressure > 150 mmHg or < 90 mmHg, or diastolic blood pressure > 90 mmHg or < 50 mmHg, or HR ≤ 40 and > 100 bpm, at Screening or Check-in; one repeat blood pressure measurement will be allowed at Screening and Check-in.
* History suggestive of esophageal (including esophageal spasm, esophagitis), gastric, or duodenal ulceration or bowel disease (including but not limited to peptic ulceration, gastrointestinal bleeding, ulcerative colitis, Crohn's disease, or irritable bowel syndrome), or a history of gastrointestinal surgery other than uncomplicated appendectomy and hernia repair.
* Inability to swallow oral medication or history of malabsorption syndrome.
* History of hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee) and in consultation with the Sponsor.
* History of major bleeding disorder (for example: hemophilia, von Willebrand disease, clotting factor deficiencies, etc).
* Participant has received a dose of an investigational drug within the past 90 days or have previously completed or withdrawn from this study or any other study investigating olpasiran or have previously received olpasiran.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-09-12 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-12-11 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected Change From Baseline in QT Corrected for Heart Rate (HR) Interval Based on the Fridericia Correction (QTcF) (ΔΔQTcF) After Olpasiran Dosing | Day 3 of Treatment Period 4 (up to approximately 9.5 weeks)

SECONDARY OUTCOMES:
Maximum Observed Concentration (Cmax) of Olpasiran | Up to 10 weeks
Time to Cmax (tmax) of Olpasiran | Up to 10 weeks
Half-life of Olpasiran (t1/2) | Up to 10 weeks
Area Under the Curve From Time 0 to the Last Quantifiable Concentration (AUClast) | Up to 10 weeks
Area Under the Curve From Time 0 to Infinity (AUCinf) | Up to 10 weeks
Change From Baseline in HR | Up to 10 weeks
Change From Baseline in QTcF | Up to 10 weeks
Change From Baseline in PR Interval | Up to 10 weeks
Change From Baseline in QRS Interval | Up to 10 weeks
Placebo-corrected Change From Baseline in HR | Up to 10 weeks
Placebo-corrected Change From Baseline in PR Interval | Up to 10 weeks
Placebo-corrected Change From Baseline in QRS Interval | Up to 10 weeks
Number of Participants with Categorical Outliers Related to the Following ECG parameter: QTcF, HR, PR, and QRS | Up to 10 weeks
Frequency of Treatment-emergent Changes in Electrocardiogram (ECG) Morphology | Up to 10 weeks
ΔΔQTcF After Moxifloxacin Dosing | Up to 10 weeks
Number of Participants With Treatment-emergent Adverse Events | Up to 10 weeks
Number of Participants With Treatment-emergent Serious Adverse Events | Up to 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (1):
- Fortrea Clinical Research Unit Limited - Leeds, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com